CLINICAL TRIAL: NCT05890170
Title: Patient-reported Outcome Measures After Implant Placement With Contour Augmentation Procedure
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Principal Investigator, Emilio Couso, Associate professor, and principal investigator, University of Bern
Other Study IDs: 2023-00754
Record Dates: First submitted 2023-05-16; First posted 2023-06-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-07

CONDITIONS: Tooth Loss; Bone Graft; Complications; Patient Satisfaction; Patient Acceptance of Health Care
MeSH Terms: conditions — Tooth Loss; Patient Satisfaction; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Short-term: Patients treated at the Department of Oral Surgery and Stomatology at the University of Bern will be potentially be recruited. Patients treated with a dental implant with contour augmentation procedure and required post-operative follow-ups as standard of care (short-term group) will be invited to participate in this study. Patients who expressed an interest to participate in this study at the clinical/phone screening examination, would be informed of the purpose and timeline of the study. All potential subjects will be required to read, understand, and sign the consent form, which included a thorough explanation of the study design, as well as expected benefits and possible risks of participating in the study without limit of time.
  Patients would received questionnaires. Data from questionnaires would be extracted by an independent investigator. Different variables would be included: 1) age, sex, systemic factors, date of the procedure; location and extension of the procedure...
  Interventions: Other: Patient Reported Outcomes Measures
- Mid-term: Patients treated at the Department of Oral Surgery and Stomatology at the University of Bern will be potentially be recruited. Patients treated with a dental implant with contour augmentation procedure done 1 to 5 years ago (mid-term group) will be invited to participate in this study. Patients who expressed an interest to participate in this study at the clinical/phone screening examination, would be informed of the purpose and timeline of the study. All potential subjects will be required to read, understand, and sign the consent form, which included a thorough explanation of the study design, as well as expected benefits and possible risks of participating in the study without limit of time.
  Patients would received questionnaires. Data from questionnaires would be extracted by an independent investigator. Different variables would be included: 1) age, sex, systemic factors, date of the procedure; location and extension of the procedure...
  Interventions: Other: Patient Reported Outcomes Measures
- Long-term: Patients treated at the Department of Oral Surgery and Stomatology at the University of Bern will be potentially be recruited. Patients treated with a dental implant with contour augmentation procedure done >5 years ago (mid-term group) will be invited to participate in this study. Patients who expressed an interest to participate in this study at the clinical/phone screening examination, would be informed of the purpose and timeline of the study. All potential subjects will be required to read, understand, and sign the consent form, which included a thorough explanation of the study design, as well as expected benefits and possible risks of participating in the study without limit of time.
  Patients would received questionnaires. Data from questionnaires would be extracted by an independent investigator. Different variables would be included: 1) age, sex, systemic factors, date of the procedure; location and extension of the procedure...
  Interventions: Other: Patient Reported Outcomes Measures

INTERVENTIONS:
Other: Patient Reported Outcomes Measures — Questionnaires and information extracted from the medical records would be collected.

SUMMARY:
Maintaining the general health and well-being of patients is the main goal of dental therapy. However, tooth extraction is indicated when teeth cannot be maintained in a status compatible with health, adequate esthetics, function, and/or for strategic reasons. A variable degree of alveolar ridge atrophy related to bone resorption is initiated immediately after removal of a tooth due to the local physiologic remodeling and the inflammatory response. Ridge resorption is more accentuated in the horizontal dimension, followed by the vertical mid-facial and vertical mid-lingual in non-molar and molar teeth. Among local periodontal phenotypic characteristics, facial bone thickness at the time of tooth extraction seems to be strongly associated with the extent of alveolar bone resorption.

Dental implants have increased in popularity due to their unique ability to replace teeth. During the planning phase of implant therapy, one of the main parameters assessed is the amount of residual alveolar ridge. Therefore, when tooth replacement therapy via dental implant is considered, adequate management of the site is critical to predictably preserve or reconstruct the architecture of the alveolar ridge, particularly in the anterior aesthetic zone, where its structure play a crucial role in the maintenance of function, health and esthetics. Generally, with appropriate treatment planning and execution, the adequate primary mechanical stability of the dental implant is achieved. However, bone and/or soft tissue augmentation procedures could be needed for the adequate management of deficient edentulous ridges at the time of implant placement, and these types of treatments could considerably increase the risk of morbidity, treatment expenses, and length of treatment time. Nevertheless, Implant placement with additional bone contour augmentation therapies have shown their effectiveness in the short-, mid- and long-term in contemporary dental practice.

However, to the present date, there is no information available in the literature regarding patient-reported outcome measures in patients that received tooth replacement therapy via dental implants with additional contour bone augmentation in the short-, mid- and long-term.

DETAILED DESCRIPTION:
This study is designed as a serial cross-sectional study. Subjects who had undergone an implant placement procedure involving bone contour augmentation procedure via GBR in the anterior aesthetic zone at the University of Bern School of Dental Medicine, Switzerland will be screened and invited for a survey. During the recall exams, patient-reported outcomes will be obtained utilizing standardized questionnaires. These outcome measures will enable us to compile short-, mid-, and long-term data about the patient-reported outcomes measures of tooth replacement therapy with dental implants and additional bone contour augmentation procedure and establish possible correlation with patient (i.e., age, sex, systemic diseases) and surgical-related factors (i.e., location and extension of the procedure, needed for vertical releasing incisions, previous management of the extraction site, etc).

The findings of this study could bring a valuable perspective on the replacement of missing teeth with dental implants and contour augmentation procedures and would provide clinicians and researchers novel knowledge to guide the clinical decision-making process.

Project population, inclusion and exclusion criteria Subjects who had undergone implant placement procedure involving bone contour augmentation procedure via Guided Bone Regeneration in the anterior esthetic zone at the University of Bern School of Dental Medicine, Switzerland will be screened and invited for a survey. The inclusion criteria are: 1) previous information on the bone augmentation procedure; 2) patients willing to provide an informed consent and attend the study, and 3) absence of any further surgical procedure involving the area of interest. The exclusion criteria are: 1) patients that would not remember where the surgical procedure was performed; 2) unwilling or unable to sign the informed consent. Besides them, and taking into consideration that no further interventions are provided in this study, no further exclusion criteria are defined.

Patients who expressed an interest to participate in this study at the clinical screening examination, would be informed of the purpose and timeline of the study. All potential subjects will be required to read, understand, and sign the consent form, which included a thorough explanation of the study design, as well as expected benefits and possible risks of participating in the study.

The initial recruitment of patients would be based on their confirmation of recalling the implant placement surgery involving the bone contour augmentation procedure via GBR, its purpose, and the area of the oral cavity where the procedure was performed. In the short-term group the patients would be followed at 1-week, 2-weeks, one and three months after surgery. Mid-term would-be patients that had the procedure performed between one up to 5 years. Long-term group would be patients that had the procedure performed from 5 years up to 20 years.

Recruitment, screening and informed consent procedure Patients treated at the Department of Oral Surgery and Stomatology at the University of Bern will be potentially be recruited. Patients treated with a dental implant with contour augmentation procedure and required post-operative follow-ups as standard of care (short-term group), or patients that had the intervention done 1 to 5 years ago (mid-term group), or longer than 5 years ago (long-term group) will be invited to participate in this study. Patients who expressed an interest to participate in this study at the clinical/phone screening examination, would be informed of the purpose and timeline of the study. All potential subjects will be required to read, understand, and sign the consent form, which included a thorough explanation of the study design, as well as expected benefits and possible risks of participating in the study without limit of time. No monetary compensation would be provided to the participants in this study.

Study procedures Patients would received questionnaires. Data for the analyses would be extracted only from the questionnaire of patients. Subjects would be asked to mark a 100mm visual analogue scale (VAS) relative to the pain/discomfort that they are/had experienced from the procedure and satisfaction with the procedure. Patients would also been given the option to mark "I do not remember" if they do not recall the answer.

Data from questionnaires would be extracted by an independent investigator. Different variables would be included: 1) age, sex, systemic factors, date of the procedure; 2) location and extension of the procedure; 3) needed for vertical releasing incisions; 4) prescription of additional medication after the 2-week post-op appointment; 5) local anatomical factors (i.e., mid-facial keratinized mucosa width), presence of adjacent teeth; 6) status of post-operative healing; 7) complications during the healing period (i.e., flap dehiscence, necrosis, bone grafting extravasation, pain, infection); 8) operator (resident or faculty member).

The duration of the evaluation visit would take no longer than 10 minutes during the recall appointment. After this visit, in the mid-term and long-term group, no more visits will be necessary for the study outcomes. For the short-term group, during the different follow-up visits as the standard of care after this type of this procedure, the patient would receive similar questionnaires relative to the pain/discomfort and/or satisfaction. Standardized Oral Health Related Questionnaries (OHIP) would be also given to the patients. All the data collected will be encrypted in Redcap Software. The key for the enecryption will be set up and stored by a person who is not involved in the study.

Withdrawal and discontinuation Only patients that would not remember where the surgical procedure was performed or unwilling and unable to sign the informed consent will not be included in this research project. In the short-term group, if the patient during the next follow-up does not want to participate anymore in the study, would not be included in this research project

ELIGIBILITY:
Inclusion Criteria:

Subjects who had undergone or will have an implant placement procedure involving bone contour augmentation procedure via Guided Bone Regeneration in the anterior esthetic zone at the University of Bern School of Dental Medicine, Switzerland will be screened and invited for a survey. The inclusion criteria are:

* Previous information on the bone augmentation procedure
* Patients willing to provide an informed consent and attend the study
* Absence of any further surgical procedure involving the area of interest.

Exclusion Criteria:

* Patients that would not remember where the surgical procedure was performed
* Unwilling or unable to sign the informed consent.
* Besides them, and taking into consideration that no further interventions are provided in this study, no further exclusion criteria are defined.

Patients who expressed an interest to participate in this study at the clinical screening examination, would be informed of the purpose and timeline of the study. All potential subjects will be required to read, understand, and sign the consent form, which included a thorough explanation of the study design, as well as expected benefits and possible risks of participating in the study.

The initial recruitment of patients would be based on their confirmation of recalling the implant placement surgery involving the bone contour augmentation procedure via GBR, its purpose, and the area of the oral cavity where the procedure was performed. In the short-term group the patients would be followed at 1-week, 2-weeks, one and three months after surgery. Mid-term would-be patients that had the procedure performed between one up to 5 years. Long-term group would be patients that had the procedure performed from 5 years up to 20 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Department of Oral Surgery and Stomatology at the University of Bern will be potentially be recruited. Patients treated with a dental implant with contour augmentation procedure and required post-operative follow-ups as standard of care (short-term group), or patients that had the intervention done 1 to 5 years ago (mid-term group), or longer than 5 years ago (long-term group) will be invited to participate in this study. Patients who expressed an interest to participate in this study at the clinical/phone screening examination, would be informed of the purpose and timeline of the study. All potential subjects will be required to read, understand, and sign the consent form, which included a thorough explanation of the study design, as well as expected benefits and possible risks of participating in the study without limit of time. No monetary compensation would be provided to the participants in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
The percentage of willingness of the patients that are undergoing or underwent the placement of implants in the anterior esthetic area with additional bone contour augmentation procedure via GBR. | Through study completion, an average of 3 months, and one year after the procedure was completed
  Primary objective

SECONDARY OUTCOMES:
- To assess whether the presence of time have an influence on the willingness of the patient to perform this type of procedure again. | Through study completion, an average of 3 months, and one year after the procedure was completed
  Secondary objective
- To assess the influence of the other variables on the willingness of the patient to perform this type of procedure, overall patient satisfaction and discomfort. | Through study completion, an average of 3 months, and one year after the procedure was completed
  Secondary objective
- To assess the influence of the other variables on the patient reported outcomes measures after this type of procedure. | Through study completion, an average of 3 months, and one year after the procedure was completed
  Secondary objective

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral Surgery and Stomatology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Araujo MG, Lindhe J. 2005. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 32(2):212-218. 2. Avila-Ortiz G, Chambrone L, Vignoletti F. 2019. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 46 Suppl 21:195-223. 3. Avila-Ortiz G, Gonzalez-Martin O, Couso-Queiruga E, Wang HL. 2020. The peri-implant phenotype. J Periodontol. 91(3):283-288. 4. Cardaropoli G, Araujo M, Lindhe J. 2003. Dynamics of bone tissue formation in tooth extraction sites. An experimental study in dogs. J Clin Periodontol. 30(9):809-818. 5. Chapple IL, Wilson NH. 2014. Manifesto for a paradigm shift: Periodontal health for a better life. Br Dent J. 216(4):159-162. 6. Chappuis V, Engel O, Reyes M, Shahim K, Nolte LP, Buser D. 2013. Ridge alterations post-extraction in the esthetic zone: A 3d analysis with cbct. J Dent Res. 92(12 Suppl):195S-201S. 7. Clementini M, Agostinelli A, Castelluzzo W, Cugnata F, Vignoletti F, De Sanctis M. 2019. The effect of immediate implant placement on alveolar ridge preservation compared to spontaneous healing after tooth extraction: Radiographic results of a randomized controlled clinical trial. J Clin Periodontol. 46(7):776-786. 8. Couso-Queiruga E, Stuhr S, Tattan M, Chambrone L, Avila-Ortiz G. 2021. Post-extraction dimensional changes: A systematic review and meta-analysis. J Clin Periodontol. 48(1):126-144. 9. Lim G, Lin GH, Monje A, Chan HL, Wang HL. 2018. Wound healing complications following guided bone regeneration for ridge augmentation: A systematic review and meta-analysis. Int J Oral Maxillofac Implants. 33(1):41-50. 10. Chappuis V, Rahman L, Buser R, Janner SFM, Belser UC, Buser D. Effectiveness of Contour Augmentation with Guided Bone Regeneration: 10-Year Results. J Dent Res. 2018 Mar;97(3):266-274. 11. Buser D, Halbritter S, Hart C, Bornstein MM, Grütter L, Chappuis V, Belser UC. Early implant placement with simultaneous guided bone regeneration following single-tooth extraction in the esthetic zone: 12-month results of a prospective study with 20 consecutive patients. J Periodontol. 2009 Jan;80(1):152-62. 12. Buser D, Wittneben J, Bornstein MM, Grütter L, Chappuis V, Belser UC. Stability of contour augmentation and esthetic outcomes of implant-supported single crowns in the esthetic zone: 3-year results of a prospective study with early implant placement postextraction. J Periodontol. 2011 Mar;82(3):342-9. 13. Ordinance on Human Research with the Exception of Clinical trials (HRO) https://www.admin.ch/opc/en/classified-compilation/20121177/index.html 14. Human Research Act (HRA) http://www.admin.ch/opc/en/classified-compilation/20121176/201401010000/810.305.pdf 15. Declaration of Helsinki (https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects ) 16. STROBE statement (http://www.jclinepi.com/article/S0895-4356(07)00436-2/pdf)